CLINICAL TRIAL: NCT04186143
Title: Effects of Closed and Open Kinetic Chain Exercises on Pain, Muscles Strength, Function, and Quality of Life In Patients With Knee Osteoarthritis In Patients With Knee Osteoarthritis
Brief Title: Effects of Closed and Open Kinetic Chain Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019900
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Care Provider
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental-Study Group (Experimental): In addition to the conservative treatment of the control group, closed cinetic chain exercises were applied for 12 weeks.
  Interventions: Other: Closed Cinetic Chain Exercises
- Active Comparator (Active Comparator): In addition to the conservative treatment of the control group, opened cinetic chain exercises were applied for 12 weeks.
  Interventions: Other: Open Kinetic Chain Exercises
- Control Group (Other): Conservative treatment was applied for 12 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Closed Cinetic Chain Exercises — Sit to stand, mini squat, anterior lunge, step up exercises are performed as Closed Cinetic Chain Exercises.
  Arms: Experimental-Study Group
Other: Open Kinetic Chain Exercises — Isometric quadriceps, isotonic quadriceps, hip extension and hip adduction exercises are performed as Open Kinetic Chain Exercises.
  Arms: Active Comparator
Other: Control Group — Control Group was followed up by conservative treatment and home program for 12 weeks and they were asked to apply the home program three days in a week. Exercise brochure was handed out for home program. Quadriceps strength and harmstring stretch exercises were applied.
  Arms: Control Group

SUMMARY:
Osteoarthritis (OA) is a heterogeneous pathology characterized by focal cartilage degeneration and the formation of new bone around the subchondral bone and joint, which is the disruption of balance between the processes of destruction and repair in subchondral area. Knee OA is a considerable cause of disability and is present in 2-3% of all disability causes. Exercises are more noticeable than other methods because they are an easy method, low cost and long-lasting. To the best of our knowledge, the studies based on this topic are scarce. Therefore, the aim of this study was to compare the effects of open and closed kinetic chain exercises on pain, functional level, quality of life and muscle strength in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a heterogeneous pathology characterized by degeneration of the posterior focal cartilage and the formation of new bone around the subchondral bone and joint, which is the disruption of the balance between the processes of destruction and repair of the joint cartilage and subchondral region. Radiologically, OA was reported in the majority of people over 65 years old and in 80% of those over 75 years old. OA is the most common joint disease in the world. Knee OA is an important health problem due to pain, functional disability and reduced quality of life in patients. Studies have shown that knee OA is associated with inadequacy and pain associated with decreased quadriceps muscle strength. Strengthening education has been shown to have positive effects on OA.

Knee OA is a significant disability cause and is present in 3% of all disability causes. OA causes disability and consequent labor loss and economic loss. Therefore, OA therapy gains importance. OA therapy is classified under three headings as pharmacological methods, non-pharmacological methods and surgical methods. In non-pharmacological methods, there are a number of studies showing the effectiveness of exercise in particular. Because it is an easy method, the cost is low and it is applicable for a long time, the exercises are more important than other methods. The literature on exercise programs with optimal gains for knee osteoarthritis has not yet been established, with numerous studies reporting the importance of different types of exercise for the treatment of knee OA in the literature. Open kinetic chain exercises are frequently used to strengthen the quadriceps muscle. Closed kinetic chain exercises have been shown to increase muscle strength and improve proprioceptive function by activating more muscle spindle and joint proprioceptors. In literature, there are researches that compare closed and open kinetic chain exercises. However, these studies mostly focus on exercises after anterior cruciate ligament reconstruction. The aim of this study was to compare the effects of open and closed kinetic chain exercises on pain, functional level, quality of life and muscle strength in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* the presence of knee osteoarthritis Grade 2 and Grade 3 based on Kellgren Lawrence Classification,
* volunteering to participate in the study.

Exclusion Criteria:

* the presence of active synovitis,
* participation physiotherapy program in the last 6 months,
* systemic and cardiovascular diseases,
* neurological and orthopedic problems affecting walking and standing,
* lower extremity surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (Pain) | 12 weeks
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. The 11-point numeric scale ranges from '0' representing no pain to '10' representing pain as bad as you can imagine or worst pain imaginable.

SECONDARY OUTCOMES:
The WOMAC Index (Functional Level) | 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) was used for functional level of participants. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright; Stiffness (2 items): after first waking and later in the day; Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Biodex System Pro 4 Isokinetic Strength Dynamometer (Muscle Strength) | 12 weeks
  Muscle strength of participants were assessed with this device. Five repeated isokinetic muscle strength tests was performed at 90º / s angular velocity in order to determine the maximal muscle strength of the muscles of the lower limb M. Quadriceps femoris and Hamstring group.
Biodex System Pro 4 Isokinetic Strength Dynamometer (Muscle Strength) | 12 weeks
  Muscle strength of participants were assessed with this device. Five repeated isokinetic muscle strength tests was performed at 120º / s angular velocity in order to determine the maximal muscle strength of the muscles of the lower limb M. Quadriceps femoris and Hamstring group.
Biodex System Pro 4 Isokinetic Strength Dynamometer (Muscle Strength) | 12 weeks
  Muscle strength of participants were assessed with this device. Five repeated isokinetic muscle strength tests was performed at 180º / s angular velocity in order to determine the maximal muscle strength of the muscles of the lower limb M. Quadriceps femoris and Hamstring group.
36-Item Short Form Survey (SF-36) (Quality of Life) | 12 weeks
  The Short Form 36 (SF-36) was standardized in 1990 as a self-report measure of functional health and well-being. Version 2.0 was published in 1996 (SF-36v2), with copyright and trademark privileges belonging to the Medical Outcomes Trust, Health Assessment Lab, and QualityMetric Incorporated. The SF-36 was designed to be a brief yet comprehensive measure of general health status. Likert scales and yes/no options are used to assess function and well-being on this 36-item questionnaire. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales. The SF-36 has been translated into more than 40 languages.

CONTACTS AND LOCATIONS:
Locations (1):
- Caner KARARTI, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Heywood S, McClelland J, Geigle P, Rahmann A, Villalta E, Mentiplay B, Clark R. Force during functional exercises on land and in water in older adults with and without knee osteoarthritis: Implications for rehabilitation. Knee. 2019 Jan;26(1):61-72. doi: 10.1016/j.knee.2018.11.003. Epub 2019 Jan 2. PMID 30611642
- [Result] Olagbegi OM, Adegoke BO, Odole AC. Effectiveness of three modes of kinetic-chain exercises on quadriceps muscle strength and thigh girth among individuals with knee osteoarthritis. Arch Physiother. 2017 Jul 19;7:9. doi: 10.1186/s40945-017-0036-6. eCollection 2017. PMID 29340203
- [Result] Resende RA, Kirkwood RN, Deluzio KJ, Morton AM, Fonseca ST. Mild leg length discrepancy affects lower limbs, pelvis and trunk biomechanics of individuals with knee osteoarthritis during gait. Clin Biomech (Bristol). 2016 Oct;38:1-7. doi: 10.1016/j.clinbiomech.2016.08.001. Epub 2016 Aug 3. PMID 27509479